CLINICAL TRIAL: NCT05349383
Title: Evaluation of Reporting of Antibody-Drug Conjugate Associated Sepsis-related Toxicities Using International Pharmacovigilance Database
Brief Title: Evaluation of Reporting of Antibody-Drug Conjugate Associated Sepsis-related Toxicities
Status: Completed | Type: Observational
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Miao Yan, PhD, Associate Professor, Central South University, Central South University
Other Study IDs: CSU20220499
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Sepsis (SMQ); Opportunistic Infections; Agranulocytosis
MeSH Terms: conditions — Sepsis; Opportunistic Infections; Agranulocytosis | interventions — Immunoconjugates; Antineoplastic Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Antibody-Drug Conjugate (ADC): Sepsis-related toxicities induced by antibody-drug conjugate(ADC). Case reported in the FDA Adverse Event Reporting System (FAERS) of Sepsis-related toxicities of patient treated by ADC, with a chronology compatible with the drug toxicity Intervention: Drug: ADC
  Interventions: Drug: Antibody-Drug Conjugate
- Common cancer drug therapies other than ADC: Sepsis-related toxicities induced by Common cancer drug therapies other than ADC.
  Case reported in the FDA Adverse Event Reporting System (FAERS) of Sepsis-related toxicities of patient treated by Common cancer drug therapies other than ADC, with a chronology compatible with the drug toxicity
  Intervention:
  Drug: Chemotherapy, targeted therapy, immunotherapy and so on.
  Interventions: Drug: Antineoplastic and immunomodulating agents other than Antibody-Drug Conjugate

INTERVENTIONS:
Drug: Antibody-Drug Conjugate — Compared the case reporting of sepsis-related toxicities among ADC and other common cancer drug therapies.
  ADC:including Gemtuzumab Ozogamicin, Trastuzumab Emtansine, Inotuzumab Ozogamicin, Enfortumab vedotin, Trastuzumab deruxtecan, Sacituzumab govitecan, Brentuximab Vedotin, Moxetumomab pasudotox, Polatuzumab Vedotin, Belantamab Mafodotin, loncastuximab tesirine and Tisotumab vedotin.
  Groups: Antibody-Drug Conjugate (ADC)
Drug: Antineoplastic and immunomodulating agents other than Antibody-Drug Conjugate — We would like to include other common cancer drug therapies such as chemotherapy, targeted therapy, immunotherapy and so on as a comparator group.
  Groups: Common cancer drug therapies other than ADC

SUMMARY:
Although antibody-drug conjugate(ADC) has proved effective in treating many cancers, few patients receiving ADC may experience rare but life-threatening sepsis-related toxicities such as sepsis and septic shock. Today, data about sepsis/septic shock are scarce.

The objective was to investigate reports of sepsis/septic shock adverse events related to ADC, including Gemtuzumab Ozogamicin, Trastuzumab Emtansine, Inotuzumab Ozogamicin, Enfortumab vedotin, Trastuzumab deruxtecan, Sacituzumab govitecan, Brentuximab Vedotin, Moxetumomab pasudotox, Polatuzumab Vedotin, Belantamab Mafodotin, loncastuximab tesirine and Tisotumab vedotin using international pharmacovigilance databases such as the FDA Adverse Event Reporting System (FAERS).

DETAILED DESCRIPTION:
Here, investigators use international pharmacovigilance databases such as the FDA Adverse Event Reporting System (FAERS) of individual safety case reports, to identify cases of sepsis-related toxicities related to ADC.

ELIGIBILITY:
Inclusion Criteria:

Case reported in the FDA Adverse Event Reporting System (FAERS) or other international pharmacovigilance database of individual safety case reports to 12/31/2022 Adverse event reported were included the report with MedDRA terms: Sepsis(SMQ), agranulocytosis(SMQ), Opportunistic infections (SMQ).

Patients treated with ADC included: Gemtuzumab Ozogamicin, Trastuzumab Emtansine, Inotuzumab Ozogamicin, Enfortumab vedotin, Trastuzumab deruxtecan, Sacituzumab govitecan, Brentuximab Vedotin, Moxetumomab pasudotox, Polatuzumab Vedotin, Belantamab Mafodotin, loncastuximab tesirine and Tisotumab vedotin. Other cancer patients received common drug therapies such as chemotherapy, targeted therapy or immunotherapy would also be included as a comparator.

Exclusion Criteria:

Chronology not compatible between ADC and adverse event (sepsis-related toxicities)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patients treated with antibody-drug conjugate and experiencing sepsis-related toxicities.
Sampling Method: Non-Probability Sample
Enrollment: 24618 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Sepsis-related toxicity of antibody-drug conjugate. | Case reported in the FDA Adverse Event Reporting System (FAERS) and other international pharmacovigilance database of individual safety case reports to 12/31/2022
  Identification and report of the sepsis-related toxicity of ADC. The research includes the report with MedDRA terms: Sepsis(SMQ), agranulocytosis(SMQ), Opportunistic infections (SMQ). Drugs investigated are ADC: Gemtuzumab Ozogamicin, Trastuzumab Emtansine, Inotuzumab Ozogamicin, Enfortumab vedotin, Trastuzumab deruxtecan, Sacituzumab govitecan, Brentuximab Vedotin, Moxetumomab pasudotox, Polatuzumab Vedotin, Belantamab Mafodotin, loncastuximab tesirine and Tisotumab vedotin.

SECONDARY OUTCOMES:
Causality assessment of reported cardiovascular events according to the WHO system | Case reported in the FDA Adverse Event Reporting System (FAERS) and other international pharmacovigilance database of individual safety case reports to 12/31/2022
Description of the type of sepsis-related toxicities depending on the category of ADC | Case reported in the FDA Adverse Event Reporting System (FAERS) and other international pharmacovigilance database of individual safety case reports to 12/31/2022
Description of the drug-drug interactions associated with sepsis-related adverse events | Case reported in the FDA Adverse Event Reporting System (FAERS) and other international pharmacovigilance database of individual safety case reports to 12/31/2022
Description of the population of patients having a sepsis-related adverse events | Case reported in the FDA Adverse Event Reporting System (FAERS) and other international pharmacovigilance database of individual safety case reports to 12/31/2022
Description of the pathologies (cancer) for which the incriminated drugs have been prescribed | Case reported in the FDA Adverse Event Reporting System (FAERS) and other international pharmacovigilance database of individual safety case reports to 12/31/2022

CONTACTS AND LOCATIONS:
Locations (1):
- Central South University, Changsha, Hunan, China